CLINICAL TRIAL: NCT01989897
Title: Effect of HSA or Saline Diluent on Immunotherapy Extract Stability as Determined by Graded ID Skin Tests
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Funding for the trial was lost so study was ended. No participants were enrolled.
Sponsor: Bryan Martin, DO (Other)
Collaborators: American College of Allergy, Asthma and Immunology (Other)
Responsible Party: Sponsor-Investigator, Bryan Martin, DO, DO, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: 2012H0217
Record Dates: First submitted 2013-06-11; First posted 2013-11-21 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Allergic Rhinitis
Keywords: diluent; rhinitis; allergic
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- diluents (Experimental): Negative control = diluent, saline with HSA--phenol Positive control = saline with 1mg/ml Histamine base
  Interventions: Drug: saline with 1mg/ml Histamine base; Drug: diluent, saline with HSA--phenol

INTERVENTIONS:
Drug: saline with 1mg/ml Histamine base
Drug: diluent, saline with HSA--phenol
  Other Names: HSA 300mcg/ml (0.03%) and Saline

SUMMARY:
This is a double-blind study with respect to the diluents used, with patients known to be allergic to the specific allergen tested. Three study sites will be involved, each testing one allergen (Cat, Mite, Timothy grass pollen). Subjects who are known to be allergic to the allergen in question will be tested with serial three-fold dilutions to determine the ID 50 and relative extract potency using the method described by Turkeltaub.

DETAILED DESCRIPTION:
The specific objective of this study is to determine the stability of immunotherapy extract dilutions. Higher dilutions (lower potency) have been shown in vitro to decrease in potency over time more rapidly than less dilute preparations. The investigators hope to determine whether there is a detectable difference in skin test reaction of dilutions of three common antigens (Cat, Timothy Grass, Dust Mite). The diluents used strongly affect the strength when extract potency is tested in vitro. Therefore, the investigators expect to find a detectable difference in skin test potency based on the diluents used (Saline vs. HSA Saline [300mcg/ml]).

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects must demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.

  2. Subjects of either gender, ages 18-60 years, with a history of allergic rhinitis related to exposure to the allergen of interest.

  3. Previous positive routine skin test to the allergen to be tested: minimum 5mm wheal diameter with 10,000BAU/mL cat or minimum 5mm wheal diameter with 10,000AU/mL Dermatophagoides farinae or minimum 8mm wheal diameter with timothy 100,000BAU/mL.

  4. AND (in addition to #3) sum of erythema after SPT of at least 50mm or erythema in largest diameter of at least 30mm.

  5. Subject's skin coloring should permit evaluation of erythema. 6. Ability to stop medication that might interfere with the results of the skin prick test.

Exclusion Criteria:

- 1. Spirometry with FEV1 below 80% of predicted normal value and/or poorly controlled asthma 2. Known pregnancy 3. Patients with a history of anaphylaxis or severe allergic reactions. 4. Patients with absolute necessity of antihistamines to control their allergies 5. Patients with active and extensive atopic dermatitis. 6. Patients that take psychotropic medication. 7. General skin hyperreactivity (Negative control greater than 3 mm wheal diameter) or with known tendency for dermatographic urticaria.

8. Patients currently under allergen immunotherapy treatment or with a history of immunotherapy treatment within the last 5 years to the extract to be tested in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
to determine the stability of immunotherapy extract dilutions | The participants will be at the study site for one visit, the visit will last approximately three (3) hours. There will be one short follow-up phone call.
  Subjects who are known to be allergic to the allergen in question will be tested with serial three-fold dilutions to determine the ID 50 and relative extract potency using the method described by Turkeltaub. This will be done by measuring skin test results in mm the goal of the testing is to get an area of redness (erythema) that is approximately 50mm

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Martin, DO, Principal Investigator — Ohio State University
Locations (1):
- Martha Morehouse Medical Plaza, 2050 Kenny Rd,Suite 2200 and Suite 2600, Columbus, Ohio, United States